CLINICAL TRIAL: NCT05146154
Title: Impact of Obesity on the Pharmacokinetics of Imipenem-Relebactam in ICU Patients
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Investigator is no longer at University of Illinois
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2021-1145
Record Dates: First submitted 2021-11-13; First posted 2021-12-06 (Actual); Last update posted 2024-11-27 (Actual); Status verified 2024-11

CONDITIONS: Obesity; Critical Illness
MeSH Terms: conditions — Obesity; Critical Illness | interventions — Imipenem; Cilastatin; relebactam; imipenem, cilastatin and relebactam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pharmacokinetic cohort (Experimental): After at least 2 doses of study drug, serial blood samples will be collected from 12 non-infected, obese ICU patients to evaluate the pharmacokinetics of imipenem and relebactam in this population.
  Interventions: Drug: Imipenem/Cilastatin/Relebactam 1.25g
- Safety cohort (Experimental): After at least 2 doses of study drug, safety will be monitored closely during study drug dosing and through 72 hours after the last dose is administered in the same 12 non-infected, obese ICU patients from the PK arm
  Interventions: Drug: Imipenem/Cilastatin/Relebactam 1.25g

INTERVENTIONS:
Drug: Imipenem/Cilastatin/Relebactam 1.25g — Imipenem/cilastatin/relebactam is a combination beta-lactam/beta-lactamase inhibitor antimicrobial marketed under the brand name Recarbrio and the approved dose is 1.25g Q6h in patients with normal renal function. The individual components of this agent must be administered together and cannot be separated. Therefore, this constitutes only one intervention. Each subject will receive at least 2 doses of study drug.
  Other Names: Recarbrio

SUMMARY:
This study is an open-label, multiple-dose pharmacokinetic study of imipenem-relebactam conducted in 12 non-infected, obese ICU patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age
2. Admitted to the ICU
3. BMI ≥40 kg/m2 and/or total body weight ≥120 kg
4. Provide a signed and dated written informed consent prior to study participation

Exclusion Criteria:

1. History of significant hypersensitivity reaction or intolerance to imipenem/cilastatin or carbapenem-based agents (doripenem, ertapenem, or meropenem +/- vaborbactam)
2. History of seizures and/or receiving 1 or more anti-epileptic agent
3. Serum creatinine ≥1.5 mg/dL
4. Estimated creatinine clearance (CLCR) <60 mL/minute as determined by Cockcroft-Gault equation:
5. Actively receiving antimicrobial therapy for treatment of a confirmed or suspected infection
6. The subject has participated in a clinical trial and has received a drug or a new chemical entity within 30 days prior to the first dose of study medication
7. Positive serum pregnancy test (for women of childbearing potential)
8. Currently breast feeding
9. Has previously participated in this study
10. Concomitant use of valproic acid or divalproex sodium
11. Any other condition that may make the patient unsuitable for the study in the judgement of the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-06-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of imipenem and relebactam | 6 months
  Peak Plasma Concentration (Cmax)
Pharmacokinetic parameters of imipenem and relebactam | 6 months
  Area under the plasma concentration versus time curve (AUC)
Pharmacokinetic parameters of imipenem and relebactam | 6 months
  Total body clearance (CLt)
Pharmacokinetic parameters of imipenem and relebactam | 6 months
  Apparent volume of distribution (Vd)

SECONDARY OUTCOMES:
Safety of imipenem and relebactam | 6 months
  Monitoring for adverse drug events

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No